CLINICAL TRIAL: NCT03146624
Title: Evaluation of Patients Satisfaction of Attachment Retained Versus Clasp Retained Obturators in Unilateral Total Maxillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sharaf Mohamed Yahia, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201512
Record Dates: First submitted 2017-05-04; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Tumour
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- attachment (Experimental): attachment retained obturator
  Interventions: Other: attachment retained obturator
- clasp (Active Comparator): clasp retained obturator
  Interventions: Other: clasp retained obturator

INTERVENTIONS:
Other: attachment retained obturator — obturator which retained by attachment
  Other Names: obturator with attachment
  Arms: attachment
Other: clasp retained obturator — obturator which retained by clasp
  Other Names: obturator with clasp
  Arms: clasp

SUMMARY:
OBJECTIVE to evaluate patients satisfaction of obturator with attachment versus conventional obturator in treatment of unilateral maxillectomy .

DETAILED DESCRIPTION:
Fourteen patients were selected according to the following criteria : patients having sufficient number of natural teeth(class I and \or class IV Aramany classification)not less than five teeth, intact soft palate , sufficient mouth opening , not exposed to radiotherapy or chemotherapy. Patients were divided into two equal groups, each of seven patients: patients of group I(Comparator) received a clasp retained obturator, while patients of group II(Intervention) received an attachment-retained obturator (RCT). The design of the definitive obturator for group I included double Aker's clasp on the first , second premolars and molars with alternating buccal and lingual retention, palatal plate as a major connector and a meshwork extension at the defect side. For group II, crown preparation of all the remaining abutments was done. Then, in the wax pattern, a lingual guiding plane was prepared and two OT Vertical attachments were attached mesial to the most anterior abutment and palatal to the second premolar and first molar . Construction of the splinted crowns were completed and the final impression was made with the splinted crowns in place to be picked up into the impression. After final try-in of the obturator, construction of the definitive obturator was completed with a hard resin hollowed obturator bulb, functional relining with soft silicone liner for both groups.

Evaluation included patient satisfaction (primary outcome)where Two scales were followed in this study which are"The Obturator Functioning Scale" and " The European Organization for Research and Treatment of Cancer Head and Neck 35"

ELIGIBILITY:
Inclusion Criteria:

1. - patients with sufficient number of natural teeth(class I and \or class IV Aramany classification),
2. - intact soft palate, 3- the mouth opening is not less than 25 mm .

Exclusion Criteria:

1- patients are exposed to radiotherapy or chemotherapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-02-21 (Actual); Study Completion 2017-03-28 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | 1 month
  questionnaires"The Obturator Functioning Scale"
patient satisfaction | 1 month
  questionnaires " The European Organization for Research and Treatment of Cancer Head and Neck 35"

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Yahia Sharaf, Cairo, Egypt